CLINICAL TRIAL: NCT04350021
Title: Effect of Low Dose Metronomic Chemotherapy in Metastatic Breast Cancer - a Two Step Study With a Retrospective Analyses Followed by a Translational Phase II Study
Brief Title: Effect of Low Dose Metronomic Chemotherapy in Metastatic Breast Cancer
Acronym: METRO
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-09-20 Version 1.2
Record Dates: First submitted 2019-12-20; First posted 2020-04-16 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer Metastatic; Chemotherapy Effect
MeSH Terms: interventions — Capecitabine; Cyclophosphamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Capecitabine, Cyclophosphamide — Capecitabine 500 mg times three, Cyclophosphamide 50 mg once daily

SUMMARY:
Low dose metronomic chemotherapy (LDMC) in patients with metastatic breast cancer (MBC) is used as a palliative regiment with the aim to prolong and improve quality of life. The effect of LDMC is not fully elucidated. The aim is to evaluate the effect of LDMC with Capecitabine and Cyclophosphamide (CX) and to discover new potential predictive markers and potential markers for monitoring treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Written and informed consent
* Breast cancer confirmed by histology
* Recurrence (local or distant) not possible to cure
* Measurable or evaluable disease
* Life expectancy of more than tree months
* ECOG (Eastern Cooperative Oncology Group) performance 0-2
* No or any lines of previous therapies for recurrent disease.
* Adequate contraception for patients of Child bearing age.

Exclusion Criteria:

* Clinically significant cardiovascular disease
* Non healing wound, Active peptic ulcer or bone fracture
* Evidence of any other disease that puts the patient at high risk for treatment-related complications

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Overall response rates | From baseline until three months after last dose.
  Radiological and Clinical evaluation
Clinical benefit defined as the proportion of patients with CR(complete respons) or PR(partial respons) and patients with stable disease for 24 weeks or more. | 24 weeks
  Complete response and Partial response

SECONDARY OUTCOMES:
Progression free survival | From baseline until three months after last dose.
  Radiological and Clinical evaluation
Overall survival | From baseline until death of any course assesed up to one year.
  Death
Tolerance and safety assessment | From baseline until three months after last dose.
  Clinical evaluation
Health-related quality of life | From baseline until three months after last dose.
  EORTC-QLQ (Quality of Life Questionnaire)-30
Evaluation of molecular characteristics in ctDNA (circulating tumor) defined as mutational changes. | From baseline until the date of first documented progression or date of death from any cause, whichever came first.
  Blood sample
Evaluation of CA (cancer associated antigen) 15-3 in relation to treatment effect | From baseline until the date of first documented progression or date of death from any cause, whichever came first.
  Blood sample
Evaluation of immune deficiency panel markers defined as changes in immune cell composition | From baseline until the date of first documented progression or date of death from any cause, whichever came first.
  Blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Colleoni M, Rocca A, Sandri MT, Zorzino L, Masci G, Nole F, Peruzzotti G, Robertson C, Orlando L, Cinieri S, de BF, Viale G, Goldhirsch A. Low-dose oral methotrexate and cyclophosphamide in metastatic breast cancer: antitumor activity and correlation with vascular endothelial growth factor levels. Ann Oncol. 2002 Jan;13(1):73-80. doi: 10.1093/annonc/mdf013. PMID 11863115
- [Background] Masuda N, Lee SJ, Ohtani S, Im YH, Lee ES, Yokota I, Kuroi K, Im SA, Park BW, Kim SB, Yanagita Y, Ohno S, Takao S, Aogi K, Iwata H, Jeong J, Kim A, Park KH, Sasano H, Ohashi Y, Toi M. Adjuvant Capecitabine for Breast Cancer after Preoperative Chemotherapy. N Engl J Med. 2017 Jun 1;376(22):2147-2159. doi: 10.1056/NEJMoa1612645. PMID 28564564
- [Background] Dellapasqua S, Bertolini F, Bagnardi V, Campagnoli E, Scarano E, Torrisi R, Shaked Y, Mancuso P, Goldhirsch A, Rocca A, Pietri E, Colleoni M. Metronomic cyclophosphamide and capecitabine combined with bevacizumab in advanced breast cancer. J Clin Oncol. 2008 Oct 20;26(30):4899-905. doi: 10.1200/JCO.2008.17.4789. Epub 2008 Sep 15. PMID 18794539